CLINICAL TRIAL: NCT04941742
Title: The Use of Fractionated Exhaled Nitric Oxide in the Diagnosis and Assessment of Disease Activity of Eosinophilic Esophagitis
Brief Title: The Use of Fractionated Exhaled Nitric Oxide in the Diagnosis and Assessment of Disease Activity of Eosinophilic Esophagitis (Validation Phase)
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Tu Thanh Mai, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-18-1019 (validation)
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active eosinophilic esophagitis
- Eosinophilic esophagitis in remission
- No eosinophilic esophagitis

SUMMARY:
The purpose of this study is to evaluate the relationship between fractionated exhaled nitric oxide, peripheral eosinophils, and plasma citrulline and ß-alanine in patients with eosinophilic esophagitis (EoE) compared to those without EoE.

The hypothesis is that a combination of elevated fractional exhaled nitric oxide, increased peripheral eosinophils, and elevated plasma citrulline and ß-alanine is associated with active EoE.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient, ages 5-18 years old, who will undergo esophagogastroduodenoscopy with biopsies at Children's Memorial Hermann Hospital, as part of the standard of care in the evaluation of EoE
* Signed informed consent by a parent or legal guardian
* Signed assent form by the child/adolescent subjects 7-18 years of age

Exclusion Criteria:

* Past medical history of active asthma, active allergic rhinitis, inflammatory bowel disease (IBD), parasitic infection, hay fever and any exposure to smoking (including secondhand smoke) because these disorders are known to affect the FeNO levels
* Active respiratory tract infections at the time of FeNO evaluation because this can affect the result of the FeNO as well
* Asthma questionnaire and/or Spirometry test consistent with asthma

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients will be recruited from the outpatient clinic of the Pediatric Gastroenterology Division of The University of Texas Health and Science Center at Houston.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Fractionated exhaled nitric oxide (FeNO) level | baseline (day of first endoscopy)
  The FeNO measurement will be performed using a hand-held analyzer, the NIOX MINO (Aerocrine, Sweden). During this non-invasive procedure the patient is asked to perform a 4-6 second single-breath exhalation into the NIOX MINO, which measures FeNO in 100s with an electrochemical sensor.
Fractionated exhaled nitric oxide (FeNO) level | at about 4-12 weeks (day of second endoscopy)
  The FeNO measurement will be performed using a hand-held analyzer, the NIOX MINO (Aerocrine, Sweden). During this non-invasive procedure the patient is asked to perform a 4-6 second single-breath exhalation into the NIOX MINO, which measures FeNO in 100s with an electrochemical sensor.

SECONDARY OUTCOMES:
Esophageal eosinophil counts as assessed by biopsy | baseline (day of first endoscopy)
Esophageal eosinophil counts as assessed by biopsy | at about 4-12 weeks (day of second endoscopy)
Blood eosinophil counts as assessed by complete blood count (CBC) | baseline (day of first endoscopy)
Blood eosinophil counts as assessed by complete blood count (CBC) | at about 4-12 weeks (day of second endoscopy)
Plasma beta-alanine level as assessed by high-performance liquid chromatography | baseline (day of first endoscopy)
Plasma beta-alanine level as assessed by high-performance liquid chromatography | at about 4-12 weeks (day of second endoscopy)
Plasma citrulline level as assessed by high-performance liquid chromatography | baseline (day of first endoscopy)
Plasma citrulline level as assessed by high-performance liquid chromatography | at about 4-12 weeks (day of second endoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Tu T Mai, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Josyabhatla R, Abrenica C, Mai T, Hashmi SS, Liu Y, Mosquera R, Van Arsdall M, Navarro F, Tchakarov A, Tatevian N, Wu G, Rhoads JM. Plasma Biomarkers and Fractional Exhaled Nitric Oxide in the Diagnosis of Eosinophilic Esophagitis. J Pediatr Gastroenterol Nutr. 2023 Jan 1;76(1):59-65. doi: 10.1097/MPG.0000000000003634. Epub 2022 Oct 11. PMID 36574003